CLINICAL TRIAL: NCT06020443
Title: Adherence to Lung Cancer Screening by Low-dose Thoracic CT in Haut-Rhin Department, France.
Acronym: DECANPHAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GHRMSA 1303; 2023-A00803-42 (Other: French Health Authority)
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: High-Risk Cancer; Lung Cancer
Keywords: screening; low dose chest computed tomography; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Low Dose chest CT Scan for Lung Cancer Screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a high risk of lung cancer (Other)
  Interventions: Procedure: Low Dose chest CT Scan for Lung Cancer Screening

INTERVENTIONS:
Procedure: Low Dose chest CT Scan for Lung Cancer Screening — Low dose CT scans will be performed for three years

SUMMARY:
The main objective of the study is to measure adherence to a lung cancer screening program using low-dose thoracic CT.

DETAILED DESCRIPTION:
Secondary objectives

1. To evaluate patient compliance over the entire duration of the screening program
2. To assess patient smoking cessation
3. To describe radiation doses received during CT scans
4. To identify organizational constraints for general practitioners
5. To compare stages at diagnosis before and after implementation of screening program

Conduct of research Eligible patients will be identified by general practitioners. Patients included will require a low-dose thoracic CT scan to be performed by a radiologist of their choice. Smoking cessation will be systematically proposed, and will be carried out by the general practitioner or a tobaccologist.

The radiation dose from thoracic CT scans should not exceed 100 mGy.cm Product Dose Length (i.e. < 1.5 mSv). Imaging reports will be forwarded to the general practitioner.

If the first CT scan is negative (T0): a second scan will be scheduled 1 year later (T1). If this second scan is also negative, in the absence of lung cancer risk factors other than smoking, scans will then be performed every two years. In the presence of a risk factor for lung cancer (other than tobacco), screening will remain annual.

In the event of a result classified as uncertain: a follow-up scan is scheduled at 3 months ; if the follow-up scan is negative, the next screening will be scheduled 1 year after this follow-up scan. If the screening performed 1 year later is also negative, subsequent screenings will be performed annually.

In the event of a positive result: the general practitioner will refer the patient to a pneumologist of his/her choice for further examinations; data from these additional examinations will be collected.

The screening protocol may evolve in line with recommendations issued by the French National Authority for Health (HAS).

For participants undergoing CT scan at the imaging department of Emile Muller hospital in Mulhouse (GHRMSA), a blood sample will be collected (optional) for subsequent biomarker assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 74 years
* Smoking OR having smoked (withdrawal of <15 years): ≥15 cigarettes/day for ≥25 years OR ≥10 cigarettes/day for ≥30 years
* Affiliated or beneficiary of a social security scheme
* Written informed consent

Exclusion Criteria:

* Inability to walk up two flights of stairs without stopping
* BMI > 35 kg/m²
* Recent chest CT scan < 1 year
* Personal history of lung cancer < 5 years or under treatment
* Personal history of cancer being monitored by chest CT scan
* Contraindication to lung cancer treatment or diagnostic investigations
* Current or recent respiratory symptoms immediately suggestive of lung cancer
* Pregnant or breast-feeding woman
* Person under court protection, guardianship or curatorship
* Person deprived of liberty by judicial or administrative decision.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of included patients having undergone the first screening scan | T0

SECONDARY OUTCOMES:
Rate of patients who refused to participate in the screening program | 1 year
Rate of included patients having completed CT scans at each stage of follow-up | 3 years
Number of patients newly committed to smoking cessation during the screening period | 3 years
Tobacco consumption | 3 years
Radiation doses received at each CT scan | 3 years
Organizational constraints of the screening program | before starting the study
  Organizational constraints of the screening program will be assessed on a subgroup of general practitioners by semi-structured interviews
Stage at diagnosis (TNM classification) of patients with lung cancer | 3 years
  The stages at diagnosis of patients with lung cancer included in the study will be compared with those of undetected patients (data from the Haut-Rhin Cancer Registry).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Strentz, MD, Principal Investigator — General Practioner, Colmar, France
Locations (1):
- Cabinet de médecine générale, Colmar, Haut-Rhin, France

IPD SHARING:
Plan to Share IPD: No